CLINICAL TRIAL: NCT01205854
Title: Aiming for Remission in Rheumatoid Arthritis: a Randomized Trial Examining the Benefit of Ultrasonography in a Clinical TIght Control Regimen
Brief Title: Aiming for Remission in Rheumatoid Arthritis (RA) - the ARCTIC Trial
Acronym: ARCTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Espen A. Haavardsholm (Other)
Collaborators: The Research Council of Norway (Other); Smerud Medical Research International AS (Other); Oslo University Hospital (Other); Innovest (Unknown); Abbott (Industry); UCB Nordic A/S (Industry); Pfizer (Industry); MSD Norway AS (Unknown); Roche Pharma AG (Industry); The Norwegian Rheumatism Association (Other)
Responsible Party: Sponsor-Investigator, Espen A. Haavardsholm, Post. doctoral Researcher, MD Ph.D., Diakonhjemmet Hospital
Organization: Diakonhjemmet Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIA2010-1
Record Dates: First submitted 2010-09-16; First posted 2010-09-21 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; ultrasonography; remission; imaging remission; tight control; treat to target
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional clinical and laboratory assessment (No Intervention)
- Conventional assessment plus ultrasonography (Experimental)
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — Standardized ultrasonographic assessment of 32 joints, assessed for both grey scale synovitis and power doppler signal, at each visit. Dose escalations based on DAS response in combination with change in US score. All joints with US Power Doppler signal are targets for intra articular injections.
  Arms: Conventional assessment plus ultrasonography

SUMMARY:
The ultimate goal of treatment in early rheumatoid arthritis (RA) is remission, i.e. an absence of signs and symptoms of the disease. However, the optimal way of reaching this goal is not known.

Ultrasonography (US) is an imaging modality which application is rapidly growing. It has a number of advantages over other advanced imaging techniques such as magnetic resonance imaging (MRI), including low cost, good accessibility, and ability to scan many joints in a short period of time. However, the additional benefit of using this modality in terms of patient outcomes has not been demonstrated. Thus, clarification is needed if the use of US leads to better care for RA patients.

This study will assess if the use of a treatment strategy incorporating information from ultrasonography assessment will allow for better outcomes of patients with RA, than a strategy based on clinical and laboratory assessments alone.

ELIGIBILITY:
Inclusion criteria (all):

* Male or non-pregnant, non-nursing female
* > 18 years of age and < 75 years of age
* Patients classified as having RA (according to new ACR/EULAR criteria)
* Disease duration less than 2 years (defined as time from 1st joint swelling)
* The treating rheumatologist decides the patient requires treatment with a Disease Modifying Anti-Rheumatic Drug (DMARD)
* The patient has taken no prior DMARD
* Patients able and willing to give written informed consent and comply with the requirements of the study protocol

Exclusion Criteria (any):

* Abnormal renal function (serum creatinine > 142 µmol/L in female and > 168 µmol/L in male)
* Abnormal liver function, active or recent hepatitis, cirrhosis
* Major co-morbidities like severe malignancies, severe diabetic mellitus, severe infections, uncontrollable hypertension, severe cardiovascular disease and/or severe respiratory diseases.
* Leukopenia and/or thrombocytopenia
* Inadequate birth control conception, pregnancy, and/or breastfeeding
* Indications of active tuberculosis
* Psychiatric or mental disorders, alcohol abuse or other abuse of substances, language barriers or other factors which makes adherence to the study protocol impossible

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2010-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Complete clinical Disease Activity Score (DAS) remission | 24 months
  Specifically, the primary endpoint will be the proportion of patients with all the following criteria met at the end of the study (at 24 months):
  * DAS score < 1.6 at visits 11, 12 and 13 (after 16, 20 and 24 months)
  * Absence of swollen joints at visits 11, 12 and 13 (after 16, 20 and 24 months)
  * No radiological progression between visit 11 (16 months) and visit 13 (24 months)

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) of dominant hand | 24 months
  MRIs of dominant hand are scored according to the Rheumatoid Arthritis Magnetic Resonance Imaging Score (RAMRIS) for synovitis, bone marrow edema and erosions, and Haavardsholm tenosynovitis score, as well as a novel joint space narrowing score will be applied.
American College of Rheumatology (ACR) response | 24 months
  Proportion of patients with ACR20, ACR50, ACR70 and ACR90 response.
Remission | 24 months
  Various definitions of remission will be calculated, including DAS-remission, ACR-remission, Simplified Diseases Activity Index (SDAI) remission and Clinical Disease Activity Index (CDAI) remission
European League Against Rheumatism (EULAR) response | 24 months
  EULAR good, moderate and non-response
Work performance | 24 months
  1. Absenteeism (work time missed)
  2. Presenteeism (impairment at work / reduced on-the-job effectiveness)
  3. Work productivity loss (overall work impairment / absenteeism plus presenteeism)
  4. Activity Impairment
Conventional radiography | 24 months
  Radiographs of hands (posterior/anterior) and foot (anterior/posterior) will be taken at baseline, 3, 6, 12, 16 and 24 months. The modified Sharp van der Heijde Score (vdHSS) will be calculated, including an erosion score and a joint space narrowing score.
The RA Impact of Disease (RAID) score | 24 months
  The RAID includes seven domains with the following relative weights: pain (21%), functional disability (16%), fatigue (15%), emotional well-being (12%), sleep (12%), coping (12%) and physical well-being (12%).
EuroQol-5 Dimension (EQ-5D) | 24 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.
Health Assessment Questionnaire (HAQ-PROMIS) | 24 months
  The HAQ-PROMIS is a questionnaire evaluating the physical function in patients with RA.
Medical Outcomes Study Short-Form 36-item (SF-36) | 24 months
  The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
Dual Energy X-ray Absorptiometry (DEXA) of spine and hip | 24 months
  Bone density measurements (DEXA hip and spine, both Z- and T-scores as well as bone mineral density) will be performed at baseline and after 12 and 24 months.
Disease Activity Score (DAS) | 24 months
  The DAS is a composite score that includes the Ritchie articular index (RAI), the 44- swollen joint counts (SJC-44), the Erythrocyte Sedimentation Rate (ESR) and a general health (GH) assessment on a Visual Analogue Scale (VAS).
  The DAS is calculated as follows:
  DAS = 0.54*sqrt(RAI) + 0.065*(SJC-44) + 0.33*Ln(ESR) + 0.0072*GH
Ultrasonography (synovitis) | 24 months
  36 joints and 2 tendons will be scored for both grey scale and power doppler synovitis on a 0-3 scale.
Magnetic Resonance Imaging (MRI) of dominant hand | 12 months
  MRIs of dominant hand are scored according to the Rheumatoid Arthritis Magnetic Resonance Imaging Score (RAMRIS) for synovitis, bone marrow edema and erosions, and Haavardsholm tenosynovitis score, as well as a novel joint space narrowing score will be applied.
American College of Rheumatology (ACR) response | 12 months
  Proportion of patients with ACR20, ACR50, ACR70 and ACR90 response.
European League Against Rheumatism (EULAR) response | 12 months
  EULAR good, moderate and non-response
Remission | 12 months
  Various definitions of remission will be calculated, including DAS-remission, ACR-remission, Simplified Diseases Activity Index (SDAI) remission and Clinical Disease Activity Index (CDAI) remission
Work performance | 12 months
  1. Absenteeism (work time missed)
  2. Presenteeism (impairment at work / reduced on-the-job effectiveness)
  3. Work productivity loss (overall work impairment / absenteeism plus presenteeism)
  4. Activity Impairment
Conventional radiography | 12 months
  Radiographs of hands (posterior/anterior) and foot (anterior/posterior) will be taken at baseline, 3, 6 and 12 months. The modified Sharp van der Heijde Score (vdHSS) will be calculated, including an erosion score and a joint space narrowing score.
The RA Impact of Disease (RAID) score | 12 months
  The RAID includes seven domains with the following relative weights: pain (21%), functional disability (16%), fatigue (15%), emotional well-being (12%), sleep (12%), coping (12%) and physical well-being (12%).
Health Assessment Questionnaire (HAQ-PROMIS) | 12 months
  The HAQ-PROMIS is a questionnaire evaluating the physical function in patients with RA.
Medical Outcomes Study Short-Form 36-item (SF-36) | 12 months
  The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
Dual Energy X-ray Absorptiometry (DEXA) of spine and hip | 12 months
  Bone density measurements (DEXA hip and spine, both Z- and T-scores as well as bone mineral density) will be performed at baseline and after 12 and 24 months.
Ultrasonography (synovitis) | 12 months
  36 joints and 2 tendons will be scored for both grey scale and power doppler synovitis on a 0-3 scale.
Disease Activity Score (DAS) | 12 months
  The DAS is a composite score that includes the Ritchie articular index (RAI), the 44- swollen joint counts (SJC-44), the Erythrocyte Sedimentation Rate (ESR) and a general health (GH) assessment on a Visual Analogue Scale (VAS).
  The DAS is calculated as follows:
  DAS = 0.54*sqrt(RAI) + 0.065*(SJC-44) + 0.33*Ln(ESR) + 0.0072*GH

CONTACTS AND LOCATIONS:
Overall Officials: Tore K Kvien, MD, PhD, Study Director — Diakonhjemmet Hospital AS
Locations (11):
- Norway (11):
  - Helse Bergen HF, Haukeland University Hospital, Dept. of Rheumatology, Bergen, Bergen
  - Martina Hansens Hospital AS, Sandvika, Bærum
  - Vestre Viken HF, Dept. of Rheumatology, Drammen, Drammen
  - Sykehuset Østfold HF, Dept. of Rheumatology, Moss, Fredrikstad
  - Haugesund Sanitetsforening Revmatismesykehus, Haugesund, Haugesund
  - Sørlandet Sykehus HF, Dept. of Rheumatology, Kristiansand, Kristiansand
  - Diakonhjemmet Sykehus AS, Dept. of Rheumatology, Oslo, Oslo County
  - Universitetssykehuset Nord-Norge HF, Dept. of Rheumatology, Tromsø, Tromsø
  - St Olavs Hospital HF, Dept. of Rheumatology, Trondheim, Trondheim
  - Revmatologene bendvold/Dovland, Kristiansand
  - Helse Sunnmøre HF, Dept. of Rheumatology, Ålesund, Ålesund

REFERENCES:
- [Derived] Sundin U, Aga AB, Skare O, Nordberg LB, Uhlig T, Hammer HB, van der Heijde D, Kvien TK, Lillegraven S, Haavardsholm EA; ARCTIC study group. Conventional versus ultrasound treat to target: no difference in magnetic resonance imaging inflammation or joint damage over 2 years in early rheumatoid arthritis. Rheumatology (Oxford). 2020 Sep 1;59(9):2550-2555. doi: 10.1093/rheumatology/kez674. PMID 31999341
- [Derived] Paulshus Sundlisaeter N, Olsen IC, Aga AB, Hammer HB, Uhlig T, van der Heijde D, Kvien TK, Lillegraven S, Haavardsholm EA; ARCTIC study group. Predictors of sustained remission in patients with early rheumatoid arthritis treated according to an aggressive treat-to-target protocol. Rheumatology (Oxford). 2018 Nov 1;57(11):2022-2031. doi: 10.1093/rheumatology/key202. PMID 30053199
- [Derived] Jonsson MK, Hensvold AH, Hansson M, Aga AB, Sexton J, Mathsson-Alm L, Cornillet M, Serre G, Lillegraven S, Fevang BS, Catrina AI, Haavardsholm EA. The role of anti-citrullinated protein antibody reactivities in an inception cohort of patients with rheumatoid arthritis receiving treat-to-target therapy. Arthritis Res Ther. 2018 Jul 13;20(1):146. doi: 10.1186/s13075-018-1635-7. PMID 30001740
- [Derived] Paulshus Sundlisaeter N, Aga AB, Olsen IC, Hammer HB, Uhlig T, van der Heijde D, Kvien TK, Lillegraven S, Haavardsholm EA; ARCTIC study group. Clinical and ultrasound remission after 6 months of treat-to-target therapy in early rheumatoid arthritis: associations to future good radiographic and physical outcomes. Ann Rheum Dis. 2018 Oct;77(10):1421-1425. doi: 10.1136/annrheumdis-2017-212830. Epub 2018 Jun 22. PMID 29934373
- [Derived] Nordberg LB, Lillegraven S, Aga AB, Sexton J, Lie E, Hammer HB, Olsen IC, Uhlig T, van der Heijde D, Kvien TK, Haavardsholm EA. The Impact of Ultrasound on the Use and Efficacy of Intraarticular Glucocorticoid Injections in Early Rheumatoid Arthritis: Secondary Analyses From a Randomized Trial Examining the Benefit of Ultrasound in a Clinical Tight Control Regimen. Arthritis Rheumatol. 2018 Aug;70(8):1192-1199. doi: 10.1002/art.40494. Epub 2018 Jun 29. PMID 29575737
- [Derived] Jonsson MK, Sundlisaeter NP, Nordal HH, Hammer HB, Aga AB, Olsen IC, Brokstad KA, van der Heijde D, Kvien TK, Fevang BS, Lillegraven S, Haavardsholm EA. Calprotectin as a marker of inflammation in patients with early rheumatoid arthritis. Ann Rheum Dis. 2017 Dec;76(12):2031-2037. doi: 10.1136/annrheumdis-2017-211695. Epub 2017 Aug 16. PMID 28814431
- [Derived] Aga AB, Berner Hammer H, Christoffer Olsen I, Uhlig T, Kvien TK, van der Heijde D, Fremstad H, Madland TM, Lexberg AS, Haukeland H, Rodevand E, Hoili C, Stray H, Noraas AL, Widding Hansen IJ, Bakland G, Lillegraven S, Lie E, Haavardsholm EA. Development of a feasible and responsive ultrasound inflammation score for rheumatoid arthritis through a data-driven approach. RMD Open. 2016 Dec 16;2(2):e000325. doi: 10.1136/rmdopen-2016-000325. eCollection 2016. PMID 28074154
- [Derived] Haavardsholm EA, Aga AB, Olsen IC, Lillegraven S, Hammer HB, Uhlig T, Fremstad H, Madland TM, Lexberg AS, Haukeland H, Rodevand E, Hoili C, Stray H, Noraas A, Hansen IJ, Bakland G, Nordberg LB, van der Heijde D, Kvien TK. Ultrasound in management of rheumatoid arthritis: ARCTIC randomised controlled strategy trial. BMJ. 2016 Aug 16;354:i4205. doi: 10.1136/bmj.i4205. PMID 27530741
- [Derived] Nordberg LB, Lillegraven S, Lie E, Aga AB, Olsen IC, Hammer HB, Uhlig T, Jonsson MK, van der Heijde D, Kvien TK, Haavardsholm EA; and the ARCTIC working group. Patients with seronegative RA have more inflammatory activity compared with patients with seropositive RA in an inception cohort of DMARD-naive patients classified according to the 2010 ACR/EULAR criteria. Ann Rheum Dis. 2017 Feb;76(2):341-345. doi: 10.1136/annrheumdis-2015-208873. Epub 2016 Apr 19. PMID 27094444
- [Derived] Aga AB, Hammer HB, Olsen IC, Uhlig T, Kvien TK, van der Heijde D, Fremstad H, Madland TM, Lexberg AS, Haukeland H, Rodevand E, Hoili C, Stray H, Bendvold AN, Soldal DM, Bakland G, Lie E, Haavardsholm EA. First step in the development of an ultrasound joint inflammation score for rheumatoid arthritis using a data-driven approach. Ann Rheum Dis. 2016 Aug;75(8):1444-51. doi: 10.1136/annrheumdis-2015-207572. Epub 2015 Jun 17. PMID 26085490